CLINICAL TRIAL: NCT06994728
Title: Characterization of Subthalamic Nucleus Deep Brain Stimulation Laterality on Visuospatial Attention and Correlation to Freezing of Gait in Parkinson's Disease
Brief Title: Correlation of STN-DBS Induced Visuospatial Changes and Freezing of Gait
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00136448
Record Dates: First submitted 2024-06-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic; Visuospatial/Perceptual Abilities
Keywords: Freezing of gait; Subthalamic nucleus; Visuospatial attention; Deep brain stimulation
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to 2 groups which will determine the side of stimulation that is kept on first while cognitive tests and assessments for freezing of gait are performed. Patients will then complete the same testing on the contralateral side.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Investigator will not be blinded as they will need to make adjustments to patient deep brain stimulation settings during testing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Left STN-DBS on, right STN-DBS off first (Active Comparator): STN-DBS will be turned off sequentially for each side, in this group beginning with left STN-DBS on and right STN-DBS off. This will then be followed by the corollary.
  Interventions: Device: Left STN-DBS on, right STN-DBS off first
- Right STN-DBS on, left STN-DBS off first (Active Comparator): STN-DBS will be turned off sequentially for each side, in this group beginning with right STN-DBS on and left STN-DBS off. This will then be followed by the corollary.
  Interventions: Device: Right STN-DBS on, left STN-DBS off first

INTERVENTIONS:
Device: Left STN-DBS on, right STN-DBS off first — There will not be any change to baseline DBS stimulation settings, only each side will be sequentially turned off during cognitive and freezing of gait assessments.
  Arms: Left STN-DBS on, right STN-DBS off first
Device: Right STN-DBS on, left STN-DBS off first — There will not be any change to baseline DBS stimulation settings, only each side will be sequentially turned off during cognitive and freezing of gait assessments.
  Arms: Right STN-DBS on, left STN-DBS off first

SUMMARY:
The purpose of this research is to determine how deep brain stimulation (DBS) for Parkinson's disease affects attention and visuospatial function. Additionally, this study will evaluate how deficits in visual attention are associated with freezing of gait (FOG) in Parkinson's disease. There is currently no reliable treatment for FOG and little is understood about the underlying reason this occurs. Some recent research has found that stimulating the right side of the brain seems to improve FOG. The right side of the brain is also paramount for visual attention, which is why investigators are conducting this study.

DETAILED DESCRIPTION:
FOG is a common and frequently disabling symptom of PD, affecting more than half of all PwPD. It remains a complex and incompletely understood phenomenon, with no currently approved therapies. FOG is often exacerbated during dual-tasks where attention is divided to multiple tasks. A well known method of provoking FOG by PwPD and neurologists alike is to walk through doorways or through a crowded space, regions where spatial attention is necessary. Similarly, significant visuospatial attention deficits have been found in PwPD who freeze compared to those do not. Further evidence demonstrates that the STN is part of the circuit which modulates spatial attention, and that STN-DBS has a significant impact on visuospatial attention and is notably improved with right sided stimulation. Indeed, visuospatial attention is largely considered to be predominantly lateralized to the right hemisphere. Interestingly, one study showed that right STN-DBS stimulation affecting a volume of activated tissue (VAT) connected to the right sensorimotor cortex showed a significant association with reduction in FOG. The impact of STN-DBS on visuospatial attention and the degree to which this change in attention is associated with changes in FOG has not yet been studied, and may well explain part of the pathophysiology of FOG and how to treat PwPD who freeze. The present study will build on the aforementioned research by prospectively evaluating the impact of lateralized STN-DBS stimulation on visuospatial attention in PwPD, and correlating this with change in FOG.

ELIGIBILITY:
Inclusion Criteria:

* Subjects above 18 years of age
* Subjects with freezing of gait
* Subjects with bilateral STN-DBS surgery as part of their clinical care for Parkinson's disease

Exclusion Criteria:

* Uncorrected visual or hearing impairments, as indicated by self-report
* Individuals who are pregnant or expect to become pregnant during the course of the study
* Individuals with dementia or relevant brain lesions impacting cognition or gait

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Characterize the individual impact of lateralized STN DBS stimulation on freezing of gait in Parkinson's disease | 1 hour
  Investigators hypothesize that right STN stimulation will have a significant association with reduction in freezing of gait, as measured by timed up and go task, compared to left STN stimulation and no stimulation.
Determine if there is a correlation between the change in visuospatial function due to lateralized STN DBS stimulation and change in freezing of gait (FOG) in Parkinson's disease | 1 hour
  Investigators hypothesize that right STN stimulation induced improvement in attention will be associated with improvement in FOG.

SECONDARY OUTCOMES:
Determine if there is a correlation between the change in Flanker task due to lateralized STN DBS stimulation in Parkinson's disease | 30 minutes
  Investigators hypothesize that right STN stimulation will have a significant association with change in attention, as measured by the flanker task, compared to left STN stimulation and no stimulation.
Determine if there is a correlation between the change in Go-No-Go task due to lateralized STN DBS stimulation in Parkinson's disease | 30 minutes
  Investigators hypothesize that right STN stimulation will have a significant association with change in attention, as measured by the Go-No-Go task, compared to left STN stimulation and no stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Nathan DeTurk, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No